CLINICAL TRIAL: NCT07219173
Title: A Phase 2, Multicenter, Randomized, Double-blind, 52-week Study, to Investigate the Efficacy and Safety of Brenipatide Compared With Placebo for the Treatment of Adult Participants With Uncontrolled Moderate to Severe Asthma
Brief Title: A Study to Evaluate Brenipatide Compared With Placebo in Adult Participants With Uncontrolled Moderate to Severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27744; 2025-522640-41 (EudraCT Number); J2S-MC-GZMR (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Incretin
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brenipatide Dose 1 (Experimental): Brenipatide administered subcutaneously (SC)
  Interventions: Drug: Brenipatide
- Brenipatide Dose 2 (Experimental): Brenipatide administered SC.
  Interventions: Drug: Brenipatide
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brenipatide — Administered SC
  Other Names: LY3537031
  Arms: Brenipatide Dose 1
Drug: Brenipatide — Administered SC
  Other Names: LY3537031
  Arms: Brenipatide Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of brenipatide at different dose levels compared with placebo in participants with moderate-to-severe asthma.

Study participation will last approximately 65 weeks, including screening, treatment, and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma who have received a physician-prescribed asthma controller medication for at least 12 months prior to screening visit.
* Participants must have an asthma control questionnaire-6 (ACQ-6) score of ≥1.5 on 2 out of 3 visits before randomization.
* History of 1 severe asthma exacerbation that led to systemic glucocorticoid treatment in the last 12 months prior to screening visit.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  * An established diagnosis of occupational asthma
* Known pre-existing, clinically important lung condition other than asthma, including but not limited to:

  * chronic respiratory infection
  * bronchiectasis
  * pulmonary fibrosis
  * allergic bronchopulmonary aspergillosis
  * emphysema
  * chronic bronchitis
  * eosinophilic granulomatosis with polyangiitis
  * chronic obstructive pulmonary disease, and
  * other mimics of asthma, that is, vocal cord dysfunction.
* Have a current or recent acute, active infection. For at least 30 days before screening visit and up to the randomization visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Annualized Asthma Exacerbation Rate Over 52 Weeks of Treatment | Baseline to Week 52
  To assess the asthma exacerbation rate.

SECONDARY OUTCOMES:
Change from Baseline in Pre-Bronchodilator (BD) Forced Expiratory Volume in One Second (FEV1) | Baseline, Week 52
Change from Baseline in Patient Reported Health Outcomes | Baseline, Week 52
Time to First Exacerbation | Baseline to Week 52
Change from Baseline in Weekly Mean Rescue Medication Use | Baseline, Week 52
Pharmacokinetic (PK): Average Steady State Plasma Concentration (Cavg) of Brenipatide | Baseline up to Week 52
Percentage of Participants with Treatment-emergent Anti-Drug Antibody (ADAs) | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-45 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (120):
- United States (17):
  - AMR Clinical, Tempe, Arizona
  - NewportNativeMD, Inc., Newport Beach, California
  - California Medical Research Associates, Northridge, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Asthma & Allergy Associates - Colorado Springs, Colorado Springs, Colorado
  - AMR Clinical, Doral, Florida
  - Renstar Medical Research, Ocala, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - USF Health, Tampa, Florida
  - Axis Clinical Trials - Westchester, Westchester, Illinois
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - AMR Clinical, Las Vegas, Nevada
  - Equity Medical, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Vanderbilt Asthma, Sinus and Allergy Program, Nashville, Tennessee
- Argentina (10):
  - Consultorios Médicos, Organización del Buen Ayre S.R.L., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Fundación Respirar, Buenos Aires
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires
  - Instituto de Asma, Alergia y Enfermedades Respiratorias, Corrientes
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Instituto Médico Río Cuarto, Río Cuarto
  - ABC Instituto de Diagnóstico, Rosario
  - Ibamedica, Santa Fe
- Brazil (10):
  - NewData Clinical Research - Aracaju, Aracaju
  - Private Practice - Dr. Nelson Rosário, Curitiba
  - Clinica de Pneumologia, Goiânia
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Hospital Universitário Onofre Lopes, Natal
  - Instituto Atena de Pesquisa Clinica, Natal
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Clinica de Alergia Martti Antila, Sorocaba
- Canada (11):
  - Dynamic Drug Advancement, Ajax
  - Heritage Medical Research Clinic, Calgary
  - University Of Alberta Hospital, Edmonton
  - St. Joseph's Healthcare Hamilton, Hamilton
  - Kelowna Health and Memory Centre, Kelowna
  - McGill University Health Centre, Montreal
  - IUCPQ, Québec
  - Richmond Clinical Trials, Richmond
  - C.I.C. Saint-Laurent, Saint-Laurent
  - Inspiration Research, Toronto
  - Dr. Syed Anees Medicine Professional Corporation, Windsor
- China (13):
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technolo -T, Baotou
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing
  - Shanghai General Hospital, Shanghai
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - The Second Afilliated Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- France (10):
  - Centre Hospitalier du Pays dAix - Centre Hospitalier Intercommunal Aix-Pertuis - Site d'Aix en Provence, Aix-en-Provence
  - CHRU de Brest, Brest
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Groupe Hospitalier Intercommunal Le Raincy-Montfermeil, Montfermeil
  - Hôpital Bichat - Claude-Bernard, Paris
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital Foch, Suresnes
- Germany (8):
  - KPPK Studienzentrum, Bendorf
  - Studienpraxis Berlin-Brandenburg Lennart Schaper, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen, Essen
  - IKF Pneumologie Frankfurt, Clinical Research Center, Departments: Pulmonology, Endocrinology, Cardiovascul -T, Frankfurt
  - ME Clinical Respiratory Research Hamburg, Hamburg
  - POIS Sachsen, Leipzig
  - IKF Pneumologie Mainz, Mainz
  - Dedicated Research Site FutureMeds, Offenbach
- India (10):
  - Galaxy Superspeciality Hospital, Aurangabad
  - Mahatma Gandhi Mission Medical College, Aurangabad
  - Medstar Speciality Hospital, Bangalore
  - All India Institute of Medical Sciences, Bhubaneswar
  - Aakash Healthcare Private Limited, Dwārka
  - Atmaram Child Care, Kanpur
  - All India Institute of Medical Sciences, New Delhi
  - Lifepoint Multispeciality Hospital, Pune
  - All India Institute of Medical Sciences, Raipur
  - Pandit Bhagwat Dayal Sharma Post Graduate Institute of Medical Sciences, Rohtak
- Japan (11):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Osaka Habikino Medical Center, Habikino
  - Aso Iizuka Hospital, Iizuka
  - Kagoshima University Hospital, Kagoshima
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Kameari Internal Medicine and Respiratory Clinic, Katsushika-ku
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
- Mexico (10):
  - San Peregrino Unidad de Investigación, Aguascalientes
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Instituto Jalisciense de Investigación Clínica Sa de Cv, Guadalajara
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - Centro de Desarrollo Biomedico, Mérida
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - Cicmex Centro de Investigación Clínica de México, Morelia
  - Centro de Investigacion Clinica Chapultepec, Querétaro
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (6):
  - EB Medical Research, Almere Stad
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis, Rotterdam
  - Gelre Ziekenhuizen, Zutphen
  - Isala, locatie Zwolle, Zwolle
- Poland (4):
  - Centrum Medyczne ,,All - Med'' Badania Kliniczne, Krakow
  - Diamond Clinic, Krakow
  - Alergologia Plus sp. z o.o., Poznan
  - Specjalistyczna Przychodnia Lekarska Alergo-Med Sp. z o.o, Poznan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement. URL: https://vivli.org/
URL: http://vivli.org/